CLINICAL TRIAL: NCT04964297
Title: Evaluation of Ability to Detect Bowel Gas During Laparoscopic Right Colectomy With Intracorporeal Anastomosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Need for device upgrade.
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Sentire Medical Systems (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-10022823
Record Dates: First submitted 2021-07-07; First posted 2021-07-16 (Actual); Results first posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Crohn's Disease of Large Intestine; Malignant Neoplasm of Colon
Keywords: Colon cancer, Crohn's disease, Perf-AlertTM device, Hydrogen gas(H2), gas Methane (CH4)
MeSH Terms: conditions — Crohn Disease; Colonic Neoplasms

STUDY DESIGN:
Intervention Model Description: Prospective pilot, single-center, single-arm, open-label, phase 1 investigator-initiated study to determine device ability to detect bowel gas during laparoscopic right colectomy with intracorporeal anastomosis using Perf-AlertTM gas detection system on 20 subjects into 2 Cohorts.
  Cohort 1: 10 subjects with measurement of bowel gas at 8 predetermined time points during right laparoscopic colectomy as follow:
  1. Initiation of surgery/laparoscopy start Insufflation
  2. Abdominal exploration
  3. Completion of colon mobilization
  4. Colon transection
  5. At Colotomy
  6. At Enterotomy
  7. Anastomosis completion
  8. End of surgery- after re-insufflation before closure
  Cohort 2: 10 subjects with continuous monitoring of bowel gases through the surgery. The level of H2 and CH4 gases will be noted at the 8 predetermined time points during the continuous monitoring as well.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Cohort 1: Predetermined points measurement (Other): Cohort 1: Predetermined points measurement: 10 subjects with measurement of bowel gas at 8 predetermined time points during right laparoscopic colectomy as follow:
  1. Initiation of surgery/laparoscopy start Insufflation
  2. Abdominal exploration
  3. Completion of colon mobilization
  4. Colon transection
  5. At Colotomy
  6. At Enterotomy
  7. Anastomosis completion
  8. End of surgery- after re-insufflation before closure
  Interventions: Device: Obtaining bowel gas samples
- Cohort 2: Continuous monitoring (Other): Cohort 2: Continuous monitoring: 10 subjects with continuous monitoring of bowel gases through the surgery. The level of H2 and CH4 gases will be noted at the 8 predetermined time points during the continuous monitoring as well.
  Interventions: Device: Obtaining bowel gas samples

INTERVENTIONS:
Device: Obtaining bowel gas samples — The Perf-AlertTM prototype consists of a 15" x 13" x 7" unit containing gas sensors and valves, a small box containing a one-way, ultra-low pressure pump, user controls (buttons), and software algorithms, which control the operation of the device. It is used in conjunction with a single-use, disposable kit of sterile tubing and filters used for sample collection. The sensing unit will be connected via a sterile tube/filter set to any trocar port in use during the procedure. At specific time points during surgery, a one-way valve will be opened, and the unit's pump turned on and withdrawing a small amount of gas from the abdominal cavity. The system is configured that sample collection, transport, analysis, and feedback occur in a single step such that sample collection and sensor feedback occur in real-time. A standard laptop running an analytical software program is connected to the unit to record and log sensor readings.

SUMMARY:
Undetected bowel perforation is a rare but dangerous complication of laparoscopic surgery. If the injury is not detected and treated at the time of the surgical procedure, the patient can suffer severe complications, including septic shock and eventually death. The investigator's goal is to test a novel device that can detect bowel gas leakage from perforation and alert the surgeon during the operation by evaluating the gases present in the insufflated abdomen during surgery. This study will determine the ability of the device to be attached to a standard trocar during the operation and periodically draw small samples or aliquots of gas from the abdomen to evaluate the gas and accurately detect gaseous content from the bowel. Before the device can be used to detect bowel perforations, the investigators must first ensure that it can accurately detect bowel gas in an insufflated abdomen.

DETAILED DESCRIPTION:
The goal of this study is to test a novel device that can detect bowel gas leakage from perforation and alert the surgeon during the operation by evaluating the gases present in the insufflated abdomen during surgery. During laparoscopic surgery, CO2 is inserted into the abdominal cavity in order to perform the operation. This is a dynamic process as insufflation is constant during the entire procedure to maintain constant pressure and compensate for any small leaks due to the insertion and retrieval of instruments.

This study will determine the ability of a novel device to be attached to a standard trocar during the operation and periodically draw a small amount of gas from the abdomen to evaluate the gas and accurately detect gaseous content from the bowel. Before the device can be used to detect bowel perforations, first the investigators must ensure that it can accurately detect bowel gas in an insufflated abdomen.

The Investigational device, Perf-AlertTM, consists of a 15" x 13" x 7" unit containing gas sensors and valves, a small box containing a one way, ultra-low pressure pump, user controls (buttons), and software algorithms, which control the operation of the device ( Image1). It is used in conjunction with a single-use, disposable kit consisting of sterile tubing and filters used for sample collection and transport (Image 2). The sensing unit will be connected via a sterile tube/filter set to any trocar port in use during the procedure. At specific time points during the procedure, a one-way valve will be opened and the unit's pump turned on pulling small aliquots of gas from the abdominal cavity to the sensing unit. The system's architecture is configured such that sample collection, transport, analysis, and feedback occur in a single step such that sample collection and sensor feedback occur in real-time. A standard laptop running an analytical software program is connected to the unit to record and log sensor readings. No changes to the device are anticipated during the course of the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years of age.
* Documentation of a required elective right laparoscopic hemicolectomy with intracorporeal anastomosis
* Subject signed inform consent

Exclusion Criteria:

* Less than 18 years old
* Pregnant or breastfeeding patients
* Patients undergoing emergency laparotomy for perforated right colon or trauma
* Patients with Intraabdominal abscess, peritonitis, or enteric fistula
* Patients who are on peritoneal dialysis
* Subjects do not speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-08-09 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mehraneh Jafari, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Predetermined Points Measurement: Cohort 1: Predetermined points measurement: 10 subjects with measurement of bowel gas at 8 predetermined time points during right laparoscopic colectomy as follow:
  1. Initiation of surgery/laparoscopy start Insufflation
  2. Abdominal exploration
  3. Completion of colon mobilization
  4. Colon transection
  5. At Colotomy
  6. At Enterotomy
  7. Anastomosis completion
  8. End of surgery- after re-insufflation before closure
  Obtaining bowel gas samples: The Perf-AlertTM prototype consists of a 15" x 13" x 7" unit containing gas sensors and valves, a small box containing a one-way, ultra-low pressure pump, user controls (buttons), and software algorithms, which control the operation of the device. It is used in conjunction with a single-use, disposable kit of sterile tubing and filters used for sample collection. The sensing unit will be connected via a sterile tube/filter set to any trocar port in use during the procedure. At specific time points during surgery, a one-way valve will be opened, and the unit's pump turned on and withdrawing a small amount of gas from the abdominal cavity. The system is configured that sample collection, transport, analysis, and feedback occur in a single step such that sample collection and sensor feedback occur in real-time. A standard laptop running an analytical software program is connected to the unit to record and log sensor readings.
Period: Overall Study
Arm/Group | Cohort 1: Predetermined Points Measurement | Cohort 2: Continuous Monitoring
Started | 3 | 0
Completed | 3 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Study enrollment closed prior to cohort 2 enrollment. Zero participants were enrolled in Cohort 2
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Predetermined Points Measurement | Cohort 2: Continuous Monitoring | Total
Number analyzed (Participants) | 3 | 0 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 1 |  | 1
  >=65 years | 2 |  | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.3 (10.4) |  | 68.3 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 |  | 0
  Male | 3 |  | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  | 0
  Not Hispanic or Latino | 3 |  | 3
  Unknown or Not Reported | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 1 |  | 1
  White | 2 |  | 2
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 |  | 3

OUTCOME MEASURES:

1. Primary Outcome: Methane (CH4) Gas
Description: Methane (CH4) gas measured in ppm or mg/L (parts per million or milligrams per liter (mg/L) at 8-time points
Time Frame: during surgery(from start of laparoscopy to the end of surgical procedure)
Population: Zero participants were enrolled in Cohort 2.
Measure: Mean (Standard Deviation); unit: ppm
Arm/Group | Cohort 1: Predetermined Points Measurement | Cohort 2: Continuous Monitoring
Number analyzed (Participants) | 3 | 0
ppm | 2.62 (0.27) |

2. Primary Outcome: Hydrogen (H2) Gas
Description: Hydrogen (H2) gas measured in ppm or mg/L (parts per million or milligrams per liter (mg/L) at 8-time points
Time Frame: during surgery(from start of laparoscopy to the end of surgical procedure)
Population: Zero participants were enrolled in Cohort 2.
Measure: Mean (Standard Deviation); unit: ppm
Arm/Group | Cohort 1: Predetermined Points Measurement | Cohort 2: Continuous Monitoring
Number analyzed (Participants) | 3 | 0
ppm | 20.69 (30.53) |

3. Secondary Outcome: Response Time of the Perf-AlertTM Device.
Description: The response time of the Perf-AlertTM device measured in seconds from obtaining the sample (from opening the valve to obtain sample) to first detecting a gas presence at the device electronic sensors
Time Frame: during surgery(from start of laparoscopy to the end of surgical procedure)
Population: Zero participants were enrolled in Cohort 2.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Cohort 1: Predetermined Points Measurement | Cohort 2: Continuous Monitoring
Number analyzed (Participants) | 3 | 0
seconds | 12 (20.78) |

ADVERSE EVENTS:
Time Frame: 90 days
Description: Zero participants were enrolled in Cohort 2.
Arm/Group | Cohort 1: Predetermined Points Measurement | Cohort 2: Continuous Monitoring
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/0
Other Adverse Events (participants affected / at risk) | 0/3 | 0/0

LIMITATIONS AND CAVEATS:
This study was terminated leading to small numbers of subjects enrolled and analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-06-03): https://cdn.clinicaltrials.gov/large-docs/97/NCT04964297/Prot_SAP_000.pdf